CLINICAL TRIAL: NCT02827773
Title: Improving Medication Adherence: A Pilot Study With Talking Pill Bottles
Brief Title: Improving Medication Adherence: A Study With Talking Pill Bottles
Acronym: TPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Dana-Farber Cancer Institute (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Seth Wolpin, Research Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35077-G
Record Dates: First submitted 2016-06-15; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Medication Adherence
Keywords: Literacy
MeSH Terms: conditions — Medication Adherence; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Received Talking Pill Bottles (Experimental): Patients received anti-hypertensives over 90 day period in Talking Pill Bottle which contained summary of pharmacy counselling session.
  Interventions: Other: Talking Pill Bottle
- Usual Care (No Intervention): Patients received oral summary of pharmacy counselling session.

INTERVENTIONS:
Other: Talking Pill Bottle — Made by Talking Rx
  Arms: Received Talking Pill Bottles

SUMMARY:
The aim of this research project is to compare the use of "Talking Pill Bottles" to usual care in patients who have low functional health literacy and who purchase medications for primary hypertension at a retail pharmacy with regard to:

1. feasibility of the procedures,
2. utility of the equipment,
3. medication adherence,
4. self efficacy in medication self management, and
5. blood pressure control.

DETAILED DESCRIPTION:
Introduction: Across the healthcare continuum, patients with low functional health literacy may have worse outcomes due to difficulties in following prescribed medication regimens. While reasons for non-adherence can be drawn from the intra-personal, interpersonal, and systemic perspectives; one starting point is the difficulty that patients have reading and understanding medication instructions on a prescription bottle labels. Labels can provide a vital reminder and decision support aid for patients and healthcare proxies. Yet, skills must be available for reading and understanding the labels. The investigators will utilize "Talking Pill Bottles" to record prescription medication instructions so that patients can re-play the instructions as needed in their homes. Purpose: The aim of this research project is to compare the use of "Talking Pill Bottles" to usual care in patients who have low functional health literacy and who purchase medications for primary hypertension at a retail pharmacy with regard to: a. feasibility of the procedures, b. utility of the equipment, c. medication adherence, d. self efficacy in medication self management, and e. blood pressure control. Design: This novel intervention will be tested within the context of a retail pharmacy in the Pacific Northwest. The pilot test will use a randomized trial design with two research arms. Analysis: Within-group change scores on a self efficacy measure and blood pressures will be examined with the paired t-test; between group measures will also be examined between the two treatment arms. The investigators will also track medication complexity as a potential confounder and conduct semi-structured exit interviews. Conclusion: Results will help establish the feasibility and utility of providing this technology to patients who have low functional health literacy in a retail pharmacy. The investigators will gather preliminary descriptive data along with variance and effect size measures for power estimations in a future multi-site, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Filling a prescription for hypertension treatment
* Able to understand spoken English.

Exclusion Criteria:

* Cannot understand English;
* Hearing impaired when not using hearing assistive devices
* Cognitively impaired.
* Unable to read labels with corrected vision

Min Age: 21 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure at 3 months | 90 days
  Measured by electronic blood pressure cuff at 90 days

SECONDARY OUTCOMES:
Change from Baseline Self Efficacy in Medication Self Administration at 3 months | 90 days
  Measured by using the survey instrument of same name at 90 days
Change from Baseline Medication Adherence at 3 months | 90 days
  Measured by using the survey instrument Morisky Medication Adherence Scale and also calculating Cumulative Medication Gap at 90 days based on pill counts.
Change from Baseline Medication Knowledge at 3 months | 90 days
  Measured by administering internally created survey instrument at 90 days.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lam A, Wolpin S, Nguyen J, Berry DL, Kurth A, Morisky DE. Is 60 seconds enough? Can talking pill bottles be used in the community pharmacy setting? J Am Pharm Assoc (2003). 2011 Sep-Oct;51(5):569-70. doi: 10.1331/JAPhA.2011.10096. No abstract available. PMID 21896452